CLINICAL TRIAL: NCT04293848
Title: Research of Music Therapy in the Development of Persons With Special Needs
Brief Title: Effect of Vibroacoustic Therapy on Acute Stress in University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Jiří Kantor, Principal Investigator, Palacky University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IGA_2019_004
Record Dates: First submitted 2020-01-24; First posted 2020-03-03 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Stress, Psychologic
Keywords: vibroacoustic therapy
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Sequentially numbered, opaque, sealed envelopes will be used as a mechanism for allocation concealment. The allocation sequence will be generated on a remote workplace by a specialist not participating on enrollment and assigning participants to intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music with low-sinusoidal sound (vibrations) (Experimental): Participants will listen to music and low-sinusoidal sound (vibroacoustic therapy).
  Interventions: Other: Vibroacoustic therapy
- Control Group (Placebo Comparator): Participants will listen to music alone.
  Interventions: Other: Only music (no vibrations)

INTERVENTIONS:
Other: Vibroacoustic therapy — listening to low-frequency sound of 40 Hz with biorhythmic sequential modulation combined to music
  Other Names: music with low-frequency sound treatment
  Arms: music with low-sinusoidal sound (vibrations)
Other: Only music (no vibrations) — listening to music, no vibrations
  Arms: Control Group

SUMMARY:
The goal of the planned Randomized Control Trial is to explore the effect of vibroacoustic therapy on acute stress of university students. The theoretical framework of the study is based on biopsychosocial model of stress and multimodal approach to measurement. The trial is designed as single-blinded, placebo-controlled, with participants individually randomized into two parallel-groups, including equal randomization and blocked allocation of participants. 420 participants are all full-time university students (18-30 years) and will be divided into two groups: an experimental group (receiving low vibrations combined with music) and a control group (only music without low-frequency sounds). For both groups acute stress response will be measured by spectral analysis of heart rate variability (HRV SA), galvanic skin response (GSR), salivary cortisol, standardized psychological questionnaires - visual analogue scales for stress (VAS-stress) and Perceived Stress Scales-10, Czech version (PSS-10). It is expected that the experimental group will demonstrate a lower level of stress response that will be measured by higher activity of parasympathetic activity, lower level of skin resistance, lower level of salivary cortisol and lower subjective perception of stress. If vibroacoustic therapy turns out to be effective, it can be viewed as safe, student-friendly and inexpensive prevention of stress-related health problems and promote the health of students in the course of university education.

DETAILED DESCRIPTION:
Primary objective: to explore whether application of vibroacoustic therapy has more significant effect on eliminating acute stress response in university students than music alone.

Research question: "Does the application of vibroacoustic therapy (low frequency vibration with music) show a more significant effect on decreasing an acute stress response (measured by HRV SA, GSR, salivary cortisol) and perception of stress (measured on VAS) in university students compared to listening to music without technologically modified low-vibrations?"

Participants: The recruitment of suitable research participants will be carried out among students studying at Faculty of Education at Palacky University in Olomouc, Czech Republic, provided that all inclusive criteria are met. Participants will be recruited by three researchers via mail and personal contact with students at the start of each of two semesters of one academic year. Only students with medium or high levels of acute stress will participate on the research experiment (level of stress measured by PSS-10, min. 20 points are required from participants). Recruiting process will be coordinated and overseen by a recruitment coordinator. Sequentially numbered, opaque, sealed envelopes will be used as a mechanism for allocation concealment. The allocation sequence will be generated at a remote workplace by a specialist not participating in enrollment and assignment of participants for the intervention.

It is a parallel group, two arms, superiority trial with 1.1. allocation ratio. Equal blocked randomization (with block size 8) with stratification according to the gender will be used here. The randomization scheme will determine which persons will be placed in the intervention group and the control group (placebo) The randomization will be implemented by a computerized random number generator (program Sealed Envelope).

The intervention is triple-blinded (blinded will be participants, statisticians as well as outcome measurements). Considering one-shot character of research experiment in every participant possibility of emergency unblinding has not been considered, nor systematic plans to promote participants´ retention and complete follow-up have not been created.

Research experiment: After recruitment students will be divided into the experimental or control groups by means of randomization. Experimental group will get full intervention including music with low-frequency sound. Control group will listen to the same music as planned for experimental group without the low-frequency sound in the frequency range 20-100 Hz (no vibrations). Measurements in two parallel groups will be carried out by two trained persons under supervision by a psychologist, physiological measurement experts and a research coordinator overseeing adherence to experimental protocols.

Measurements: The measurement methods consist of (1) heart rate variability spectral analysis, (2) galvanic skin response, (3) salivary cortisol, (4) Perceived Stress Scale questionnaire, (5) visual analogue scales for stress and (6) a questionnaire of own construction.

Statistical analysis: Data analysis methods will be based on statistical processing in the form of the one-way (factor Vibroacoustic/Placebo) repeated measures (factor Before/After) ANOVA. The intervention arm will be compared against the control for all primary analyses and significant differences in the responses of autonomous nervous system, salivary cortisol and the stress perception will be examined.

Hypotheses:

H1: Listening to vibroacoustic therapy recording (music with low-frequency vibrations) will stimulate higher levels of parasympathetic nervous activity compared to listening to music alone.

H2: Listening to vibroacoustic therapy recording (music with low-frequency vibrations) will stimulate lower levels of salivary cortisol compared to listening to music alone.

H3: Listening to vibroacoustic therapy recording (music with low-frequency vibrations) will stimulate lower levels of subjective perception of stress compared to listening to music alone.

ELIGIBILITY:
Inclusion Criteria:

* participants want to voluntarily participate in the study,
* they are 18-30 years old,
* they are of Czech or Slovak nationality,
* full-time students.

Exclusion Criteria:

* psychiatric diagnosis,
* neurologic disease (e.g. epilepsy, cerebral palsy) or any known contraindication of vibro-acoustic therapy such as muscle hypotonia, angina pectoris, psychotic or acute post-traumatic and bleeding,
* post-traumatic stress disorder,
* perceived pain,
* persons after sleep deprivation,
* substance abuse (caffeine, nicotine) on the day of experiment and in case of strong addictive substances (alcohol, drugs) 1 day before the experiment,
* increased physical activity on the day before the experiment,
* menstruation on the day of the experiment,
* moderate to high food intake on the day of the experiment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
subjective stress perception | 1 day
  Subjective stress perception measured by Visual Analogue Scales for Stress and Perceived Stress Scales-10, Czech version.
Spectral analysis of heart rate variability | 1 day
  Spectral analysis of heart rate variability to measure the response of autonomous nervous system response measured by VLV Lab.
Galvanic skin response | 1 day
  Galvanic skin response to measure the response of autonomous nervous system response measured by VLV Lab.
Salivary cortisol | 1 day
  Salivary cortisol to measure the level of cortisol by Salivette Cortisol.

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Kantor, PhD, Principal Investigator — Faculty of Education, Palacky University, Olomouc, Czech Republic
Locations (1):
- Faculty of Education, Palacký University Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Only a dean and dean-deputy (as trial investigators) will be allowed an access to the full dataset before their publication based on a formal request.
Supporting Information: Study Protocol
Time Frame: From July 2021 - on